CLINICAL TRIAL: NCT07349823
Title: Exploratory Study on the Treatment of Relapsed and Refractory Immune Related Diseases With WGb-0301 Injection
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Jiyan Liu, Professor, West China Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 0301-IIT-ADs
Record Dates: First submitted 2026-01-05; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Autoimmune Diseases
MeSH Terms: conditions — Autoimmune Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WGb-0301 injection, Escalation doses (Experimental)
  Interventions: Drug: WGb-0301 injection
- WGb-0301 injection, Extended doses (Experimental)
  Interventions: Drug: WGb-0301 injection

INTERVENTIONS:
Drug: WGb-0301 injection — Drug targeting CD19 based on mRNA-LNP

SUMMARY:
The exact etiology and pathogenesis of immune related diseases (such as autoimmune hepatitis, systemic lupus erythematosus, etc.) have not been fully elucidated, and are generally believed to be the result of multiple factors such as genetics, environment, and immune regulation abnormalities. The current standard treatment for immune related diseases includes corticosteroids, biologics (such as belimumab, rituximab), and immunosuppressants (such as mycophenolate mofetil, azathioprine, cyclophosphamide, etc.). Although hormones and traditional immunosuppressants can widely suppress immunity, there are risks of bone marrow suppression, liver and kidney function damage, and long-term malignant tumors. Some patients are ineffective with glucocorticoid therapy, and some patients relapse after discontinuation of medication. Although there are various treatment methods currently available, there are still many limitations to immune related diseases that aim for long-term remission, and further research and breakthroughs are urgently needed.

Research has shown that abnormal activation of B cells is one of the important mechanisms involved in the occurrence and development of immune related diseases. Therefore, therapeutic drugs targeting B cells, such as CD20 monoclonal antibodies, have been recommended by guidelines for the treatment of refractory and recurrent immune related diseases. The therapy targeting CD19, another B-cell target, has become an important research and development direction in the treatment of immune related diseases due to its ability to clear a wider range of B-cell lineages, including plasma cells and long-lived plasma cells, showing potential long-term remission effects.

The experimental drug WGb 0301 injection is a CD19 based messenger ribonucleic acid (mRNA) therapeutic drug, formed by loading mRNA encoding CD19 receptor related proteins onto lipid nanoparticles (LNP).

ELIGIBILITY:
Inclusion Criteria:

* 1. Age range of 18-70 years old (including threshold), gender not limited;
* 2. KPS score>60 points, life expectancy greater than 6 months;
* 3. Male and female patients of appropriate age must use reliable methods of contraception before entering the trial, during the research process until 30 days after discontinuation of medication; Reliable contraceptive methods will be determined by the primary researchers or designated personnel;
* 4. Those who can understand this experiment and have signed the informed consent form;
* 5. Before screening (at baseline), corresponding requirements should be met;
* 6. Diagnosed with recurrent or refractory immune related diseases, including systemic lupus erythematosus (SLE), autoimmune hepatitis, idiopathic inflammatory myopathy, scleroderma, etc.

Exclusion Criteria:

* 1. Study participants who are allergic or hypersensitive to any component of the investigational drug, including those who are allergic to messenger RNA (mRNA) vaccines or other RNA LNP products.
* 2. Merge any active infections that require antibiotic treatment and have not been controlled for at least one week prior to administration.
* 3. Accompanied by other uncontrolled malignant tumors.
* 4. History of cardiovascular disease within the first 6 months of screening: NYHA defined grade III or IV heart failure, myocardial infarction, unstable angina, uncontrolled or symptomatic atrial arrhythmias, any ventricular arrhythmias, or other clinically significant heart diseases.
* 5. New York Heart Association (NYHA) grade III-IV heart failure.
* 6. Hepatitis B surface antigen (HBsAg) and/or hepatitis B core antibody (HBcAb) positive, and hepatitis B virus (HBV) DNA positive or titer higher than the detection threshold; Individuals with positive hepatitis C virus (HCV) antibodies and HCV RNA positivity or titers above the detection threshold; Human immunodeficiency virus (HIV) antibody positive individuals; Cytomegalovirus (CMV) DNA positive or above the detection limit; Individuals who are positive for syphilis antigen or antibody.
* 7. Vaccination with attenuated live vaccine or protein subunit vaccine within 30 days prior to the first study use.
* 8. Women who are currently pregnant, breastfeeding, or planning to become pregnant.
* 9. The researchers believe that there are other situations that are not suitable for participating in this clinical study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2026-01-26 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) and its incidence rate | Within 90 days after the initial treatment
Maxmum tolerated dose (MTD) or optimal biological dose (OBD) | Through study completion, an average of 2 years

SECONDARY OUTCOMES:
Preliminary efficacy evaluation: The degree and rate of remission of biochemical indicators | Through study completion, an average of 2 years
Preliminary efficacy evaluation: The degree and rate of remission of immunological indicators | Through study completion, an average of 2 years